CLINICAL TRIAL: NCT00010439
Title: A Non-Randomized, Open-Label, Prospective, Non-Controlled, 12-Month Clinical Trial to Determine the Effects of Alendronate 35 or 70 mg/Week Depending Upon Body Weight, in Children and Adolescent With IJO
Brief Title: Phase II Study of Alendronate Sodium in Children With High-Turnover Idiopathic Juvenile Osteoporosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Deborah A Bowlby, MD., Assistant Professor, Medical University of South Carolina
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 199/15705; FD-R-001847-01 (Other Grant/Funding Number: FDA)
Record Dates: First submitted 2001-02-02; First posted 2001-02-02 (Estimated); Results first posted 2010-09-17 (Estimated); Last update posted 2010-11-08 (Estimated); Status verified 2010-10

CONDITIONS: Osteoporosis
Keywords: arthritis & connective tissue diseases; idiopathic juvenile osteoporosis; rare disease
MeSH Terms: conditions — Osteoporosis; Arthritis; Connective Tissue Diseases; Juvenile osteoporosis; Rare Diseases | interventions — Alendronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 Alendronate for 12 months (Experimental): Ten children will take alendronate 35mg or 70mg weekly depending upon the body weight for 12 months. Patients will also take calcium supplement daily.
  Interventions: Drug: Alendronate

INTERVENTIONS:
Drug: Alendronate — Pill, 35mg or 70mg weekly, depending upon the body weight for 12 months.
  Other Names: Fosamax

SUMMARY:
OBJECTIVES:

I. Determine the effects of alendronate sodium on skeletal remodeling and bone mineral density of the hip and spine in children with high-turnover idiopathic juvenile osteoporosis.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients receive oral alendronate sodium weekly for 1 year. Treatment continues in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Eligibility Criteria:

* 5-14 years of age
* Weight 20 kg or greater
* History of one or more atraumatic fracture
* Sexual development no greater than Tanner II
* Osteoporosis by DXA (Diagnosis of high-turnover osteoporosis with no underlying cause (e.g., malignancy, hyperthyroidism, hyperparathyroidism, or vitamin D intoxication)

Inclusion Criteria:

* Male and female children with a history of one or more atraumatic fractures, or evidence of one or more compression fractures on radiographs of the spine (reduction of >20%).
* Bone mineral density by DXA at 2 standard deviations (SD) below normal mean for age (Z-score at least 2 SD below normal mean at the lumbar spine or hip)
* Parental consent (and patient assent after age 12 years) to participate in the study.
* Sexual development at Tanner stage II or less (Prepubertal stage)
* Weight 20kg and more

Exclusion Criteria:

* History of severe gastritis or reflux
* Marked kyphoscoliosis or inability to sit or stand for at least 30 minutes.
* Abnormalities of the esophagus that delay emptying (e.g., strictures or achalasia)
* Hypersensitivity to bisphosphonates
* Uncorrected hypocalcemia
* History of gastric or duodenal ulcers
* Renal dysfunction as indicated by serum Creatinine greater than 1.5 mg/dL
* Liver dysfunction as indicated by serum SGPT greater than 2 times upper limit of normal for age or serum total bilirubin greater than 2.0 mg/dL
* Diagnosis of osteogenesis imperfecta (including family history) or blue sclerae or deafness
* Diagnosis of active rickets, osteomalacia, or bone alkaline phosphatase > 2 times normal for age
* Severe gastritis or reflux
* Pregnancy
* Anorexia Nervosa

  * Prior/Concurrent Therapy-
* Prior course of prednisone allowed
* No concurrent prednisone except inhaled steroids
* No concurrent high-dose glucocorticoids
* No concurrent salmon calcitonin
* No other concurrent bisphosphonates
* No concurrent long-term anti-seizure medication

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2000-09; Primary Completion 2003-10 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Bowlby, M.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Result] Key LL Jr, Ries W, Madyastha P, Reed F. Juvenile osteoporosis: recognizing the risk. J Pediatr Endocrinol Metab. 2003 May;16 Suppl 3:683-6. PMID 12795371
- See also: "Click here for more information about this study:" — http://www.musckids.com/research/fosamax_trial.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of the recruitment period: 5/3/2001 to 7/23/2002. Types of location: Out-patient clinic, Clinical and Translational Research Center (CTRC, formerly General Clinical Research Center), Medical University of South Carolina.
Groups:
- Alendronate: Ten children will take alendronate 35mg or 70mg weekly depending upon the body weight for 12 months. Patients will also take calcium supplement daily.
Period: Overall Study
Arm/Group | Alendronate
Started | 10
6 Months | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Alendronate
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years]
  Pre-Treatment (Baseline) | 9.4 (2.3)
  Post Treatment | 10.6 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Increased Bone Mineral Density
Description: Number of participants with increase in bone mineral density at Lumbar Spine and/or Hip at 12 months as compared to the bone mineral density at Lumbar Spine and/or Hip obtained before therapy (baseline values)
Time Frame: at 12 months
Population: per protocol
Measure: Number; unit: participants
Arm/Group | Alendronate
Number analyzed (Participants) | 10
participants | 10 (0.11)

2. Secondary Outcome: Participants (1) With Fractures Before and After Therapy,(2)Analysed for Average Changes From High to Near Normal Mineral Apposition Rate (MAR) After Therapy,(3)Analysed for Average Insignificant Changes in Biochemical Markers After Therapy.
Description: Participants (pts) with fractures bef.and aft.therapy; pts analysed for average changes in mineral apposition rate (MAR) (high (1.9um/day) to near normal (1.2 um/day)as revealed in bone biopsies. MAR is the distance between the two tetracycline labels (um/day). The data represent the average of 10-17 measurements of the disltance obtained by reading 2-7 individual slides of bone biopsy and pts analysed for average insignificant biochemical markers (serum bone specific alkaline phosphatase for bone formation and urinary N-telopeptide for resorption)to determine the effect of therapy.
Time Frame: Before and 12 months after treatment with alendronate
Population: Per protocol
Measure: Number; unit: participants
Arm/Group | Alendronate
Number analyzed (Participants) | 9
participants
  Participants with fractures before therapy. | 9
  Participants with fractures after therapy. | 1
  Pts average MAR near normal after therapy | 9
  Pts av biomarker change insignificant aft. therapy | 9

ADVERSE EVENTS:
Arm/Group | Alendronate
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreement with Merck: to submit a copy of any proposed abstract, manuscript and/or press release to Merck for review and comment at least 30 days prior to submission for publication or presentation.